CLINICAL TRIAL: NCT06311552
Title: Optimising CMR Scan Acquisitions for Novel Equipment/Sequences in Clinical Cardiovascular Populations.
Acronym: OPTMISE-HFpEF
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0856
Record Dates: First submitted 2024-02-29; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CMR scan on either a 1.5- or 3-Tesla scanner
  Interventions: Other: Participants will undergo a comprehensive CMR scan on either a 1.5- or 3-Tesla scanner

INTERVENTIONS:
Other: Participants will undergo a comprehensive CMR scan on either a 1.5- or 3-Tesla scanner — Participants will undergo a comprehensive CMR scan on either a 1.5- or 3-Tesla scanner

SUMMARY:
The purpose of this study is to develop robust protocols for the optimisation of novel hardware, software and exercise equipment in the magnetic resonance imaging (MRI) environment in various cohorts with cardiovascular disease (CVD) with the first study focusing on those with established heart failure with preserved ejection fraction (HFpEF) or those at risk of or with pre-HFpEF.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged >18 years
* Either a clinical diagnosis of HFpEF, be at risk of or pre- HFpEF

Exclusion Criteria:

* Absolute contraindication to MRI
* Unable to read/understand English sufficiently to provide informed consent
* Pregnancy
* Unable to consent due to lack of mental capacity
* Current cancer diagnosis and actively undergoing treatment
* Inability to exercise on the MRI ergometer
* Severe claustrophobia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Either a clinical diagnosis of HFpEF, be at risk of or pre-HFpEF
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
To develop CMR scanning protocols which acquire the highest quality images during incremental exercise using a stepper ergometer (Ergospect Cardio-stepper). | By end of study - 30/04/2023

SECONDARY OUTCOMES:
To determine the reproducibility of the exercise CMR protocols in a test-retest reproducibility sub-study | By end of study - 30/04/2023
To determine the optimal scan acquisition protocol for Magnetic Resonance Spectroscopy (MRS) both H+ and 31P using the phosphorous coil in each patient group. | By end of study - 30/04/2023
To determine the reproducibility of the MRS protocols in a test-retest reproducibility sub-study | By end of study - 30/04/2023

CONTACTS AND LOCATIONS:
Locations (1):
- Glenfield Hospital, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: No